CLINICAL TRIAL: NCT00985608
Title: Efficacy of Acetilcysteine in 'Rescue' Therapy for Helicobacter Pylori Infection. Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Giovanni Cammarota, MD, Catholic University of the Sacred Heart-Institute of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 253/09
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: H pylori; eradication therapy
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B: antibiotic treatment (control) (Active Comparator): patients receiving solely a culture-guided one-week antibiotic treatment including a PPI plus two antibiotics
  Interventions: Drug: Group B: antibiotic treatment (control)
- Group A: NCA 600mg +antibiotics (Active Comparator): NCA 600mg once a day for a week and subsequently a culture-guided one-week regimen including a PPI plus two antibiotics
  Interventions: Drug: Group A: NCA 600 mg+antibiotics

INTERVENTIONS:
Drug: Group A: NCA 600 mg+antibiotics — NCA 600mg once a day for a week and subsequently a culture-guided one-week regimen including a PPI plus two antibiotics
  Arms: Group A: NCA 600mg +antibiotics
Drug: Group B: antibiotic treatment (control) — patients receiving solely a culture-guided one-week antibiotic treatment including a PPI plus two antibiotics
  Arms: Group B: antibiotic treatment (control)

SUMMARY:
H pylori gastric infection is one of the most prevalent infectious diseases worldwide. The discovery that most upper gastrointestinal diseases are related to H pylori infection and therefore can be treated with antibiotics is an important medical advance. Currently, a first-line triple therapy based on proton pump inhibitor (PPI) or ranitidine bismuth citrate (RBC) plus two antibiotics (clarithromycin and amoxicillin or nitroimidazole) is recommended by all consensus conferences and guidelines. Even with the correct use of this drug combination, infection can not be eradicated in up to 23% of patients. Therefore, several second line therapies have been recommended. A 7 d quadruple therapy based on PPI, bismuth, tetracycline and metronidazole is the more frequently accepted. However, with second-line therapy, bacterial eradication may fail in up to 40% of cases. When H pylori eradication is strictly indicated the choice of further treatment is controversial. When available, endoscopy with culture and consequent antibiotic susceptibility testing remains the most appropriate option for patients with two eradication failures to avoid a widespread use of expensive antibiotics. The use of these drugs may also induce severe side-effects and development of H pylori resistant strains.

Resistant strains of Helicobacter pylori can display a dense biofilm with mucus and microorganisms in a coccoid shape on the mucosal surface of stomach that may have a role in determining the resistance to the antibiotic therapies. Possibly, N-acetil-cysteine (NAC) may dissolve biofilm architecture and help to eradicate resistant strains of H pylori.

DETAILED DESCRIPTION:
To evaluate the usefulness of NAC as pre-treatment attempt associated with a culture-guided antibiotic therapy as rescue therapy after multi-attempts antibiotic failure, in the first phase of the study, the effect of NAC on biofilm formation and on its demolition will be tested in vitro by adding NAC in cultured H pylori isolates from a limited number of patients (n10) with an history of at least 4 failed eradicating attempts. Two biopsy samples of gastric mucosa will be obtained during endoscopy for microbiological purpose. Specimens will be used for H pylori culture. In specimens from 5 patients, H pylori will be cultured together with NAC 2 mg, while in the other 5 cases, H pylori culture will be carried out without NAC. In these latter, after the biofilm formation, H pylori isolates will be faced with different doses of NAC (2 mg, 10 mg, and 20 mg) to observe the behavior of biofilm. In the second phase of the study, 40 patients, after at least four unsuccessful H pylori eradication attempts, will be consecutively recruited. During endoscopy, in each patient, at least 4 mucosal biopsies will be obtained from the gastric body. Two of these biopsies will be used for biofilm study at the scanning electron microscopy (SEM). The remaining biopsies will be used for H pylori culture. From culture, the in vitro antibiotic susceptibility testing together with genetic analysis of H pylori isolates will be performed. On the basis of antibiotic susceptibility testing alone, patients will then randomly assigned to receiving two different eradication schedules: Group A, patients receiving NCA 600 mg once a day for a week and subsequently a culture-guided one-week regimen including a PPI plus two antibiotics against H pylori; group B (control), patients receiving solely a culture-guided one-week antibiotic treatment including a PPI plus two antibiotics. Sensitive antibiotics will be always chosen on the basis of the more favorable minimum inhibiting concentration value. all patients will have a diary to record the side effects and symptoms during therapy. Compliance will measured by counting the tablets returned after the 7-day treatment. Patients will take a control C13 urea breath test at least two months after the end of therapy. They will be also invited to repeat endoscopic examination for monitoring biofilm persistence or absence. Finally, results obtained with the two treatment arms will be compared and evaluated also on the light of genetic analyses of H pylori isolates.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age > 18 years
* Persistent infection from Helicobacter pylori, at gastroscopy or 13C urea breath test, after at least two antibiotic unsuccessful eradication attempts

Exclusion Criteria:

* Verified allergies to the acetylcysteine or to the antibiotics to cure Helicobacter pylori
* Pregnancy, nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the usefulness of NAC as pre-treatment attempt associated with a culture-guided antibiotic therapy as rescue therapy after multi-attempts antibiotic failure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cammarota, MD, Principal Investigator — Catholic University, Institute of Internal Medicine
Locations (1):
- Institute of Internal Medicine - Catholic University, Rome, Italy